CLINICAL TRIAL: NCT02989233
Title: Impact of Three Different Education Methods on Oral Hygiene and Theoretical Knowledge of Schoolchildren
Brief Title: Impact of Three Different Education Methods on Oral Hygiene
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Umut BALLI (Other)
Responsible Party: Sponsor-Investigator, Umut BALLI, Faculty of Dentistry, Bulent Ecevit University
Organization: Bulent Ecevit University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36290600/93
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Oral Hygiene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- Brochure-Female-8/10 (Active Comparator): Female 8-10 years Theoretical Test Application Giving a brochure Bleeding on probing, plaque index and gingival index Non-surgical periodontal treatment
  Interventions: Other: Non-surgical periodontal treatment
- Brochure-Male-8/10 (Active Comparator): Male 8-10 years Theoretical Test Application Giving a brochure Bleeding on probing, plaque index and gingival index Non-surgical periodontal treatment
  Interventions: Other: Non-surgical periodontal treatment
- Model-Female-8/10 (Active Comparator): Female 8-10 years Theoretical Test Application Expression with a model Bleeding on probing, plaque index and gingival index Non-surgical periodontal treatment
  Interventions: Other: Non-surgical periodontal treatment
- Model-Male-8/10 (Active Comparator): Male 8-10 years Theoretical Test Application Expression with a model Bleeding on probing, plaque index and gingival index Non-surgical periodontal treatment
  Interventions: Other: Non-surgical periodontal treatment
- Video-Female-8/10 (Active Comparator): Female 8-10 years Theoretical Test Application Showing a video Bleeding on probing, plaque index and gingival index Non-surgical periodontal treatment
  Interventions: Other: Non-surgical periodontal treatment
- Video-Male-8/10 (Active Comparator): Male 8-10 years Theoretical Test Application Showing a video Bleeding on probing, plaque index and gingival index Non-surgical periodontal treatment
  Interventions: Other: Non-surgical periodontal treatment
- Brochure-Female-11/13 (Active Comparator): Female 11-13 years Theoretical Test Application Giving a brochure Bleeding on probing, plaque index and gingival index Non-surgical periodontal treatment
  Interventions: Other: Non-surgical periodontal treatment
- Brochure-Male-11/13 (Active Comparator): Male 11-13 years Theoretical Test Application Giving a brochure Bleeding on probing, plaque index and gingival index Non-surgical periodontal treatment
  Interventions: Other: Non-surgical periodontal treatment
- Model-Female-11/13 (Active Comparator): Female 11-13 years Theoretical Test Application Expression with a model Bleeding on probing, plaque index and gingival index Non-surgical periodontal treatment
  Interventions: Other: Non-surgical periodontal treatment
- Model-Male-11/13 (Active Comparator): Male 11-13 years Theoretical Test Application Expression with a model Bleeding on probing, plaque index and gingival index Non-surgical periodontal treatment
  Interventions: Other: Non-surgical periodontal treatment
- Video-Female-11/13 (Active Comparator): Female 11-13 years Theoretical Test Application Showing a video Bleeding on probing, plaque index and gingival index Non-surgical periodontal treatment
  Interventions: Other: Non-surgical periodontal treatment
- Video-Male-11/13 (Active Comparator): Male 11-13 years Theoretical Test Application Showing a video Bleeding on probing, plaque index and gingival index Non-surgical periodontal treatment
  Interventions: Other: Non-surgical periodontal treatment

INTERVENTIONS:
Other: Non-surgical periodontal treatment — Scaling and oral hygiene instructions with brochure, model or video

SUMMARY:
In the present study, 144 children (72 males and 72 females), whose ages ranged between 8-13, were divided into 12 equal experimental groups according to their ages and gender. They were all considered to have poor hygiene. Only one out of the three different education methods (brochure, model or video) was applied to each group. The percentage change in PI, GI, BOP and theoretical test points from the baseline to the 6th months were evaluated.

DETAILED DESCRIPTION:
Aim: The aim the present study was to evaluate the impact of three different education methods on the oral hygiene levels of school children using clinical and theoretical findings.

Methods: In the present study, 144 children (72 males and 72 females), whose ages ranged between 8-13, were divided into 12 equal experimental groups according to their ages and gender. They were all considered to have poor hygiene. Only one out of the three different education methods (brochure, model or video) was applied to each group. The percentage change in PI, GI, BOP and theoretical test points from the baseline to the 6th months were evaluated. The data was statistically analysed by using Kolmogorov-Smirnov and One-way ANOVA tests.

ELIGIBILITY:
Inclusion Criteria:

* According to the Simplified Oral Hygiene Index, the patients having the score of 2 and over were accepted.

Exclusion Criteria:

* According to the Simplified Oral Hygiene Index, the patients having the score under 2 were not included in the study

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 144 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Theoretical Test Application | Baseline and 6 months after treatment
  The changes in theoretical test scores after education

SECONDARY OUTCOMES:
Gingival index | Baseline and 6 months after treatment
  The changes in gingival index after education
Plaque index | Baseline and 6 months after treatment
  The changes in plaque index after education
Bleeding on probing | Baseline and 6 months after treatment
  The changes in bleeding on probing after education

IPD SHARING:
Plan to Share IPD: No